CLINICAL TRIAL: NCT05817435
Title: A Phase 1, Randomized, Open-label, Parallel-Group, Single-Dose, Bioequivalence Study of Efgartigimod PH20 SC Administered Via a Prefilled Syringe Versus a Vial + Syringe Presentation in Healthy Adults
Brief Title: A Phase 1 Bioequivalence Study of Efgartigimod PH20 SC Administered Via a Prefilled Syringe Versus a Vial+Syringe Presentation in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ARGX-113-2204
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Bioequivalence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efgartigimod PH20 SC - prefilled syringe (Experimental): efgartigimod PH20 SC administered by a prefilled syringe
  Interventions: Biological: efgartigimod PH20 SC as a prefilled syringe presentation
- Efgartigimod PH20 SC - vial + syringe (Active Comparator): efgartigimod PH20 SC administered by a vial + syringe
  Interventions: Biological: efgartigimod PH20 SC as a vial + syringe presentation

INTERVENTIONS:
Biological: efgartigimod PH20 SC as a prefilled syringe presentation — efgartigimod PH20 SC as a prefilled syringe presentation
  Arms: Efgartigimod PH20 SC - prefilled syringe
Biological: efgartigimod PH20 SC as a vial + syringe presentation — efgartigimod PH20 SC as a vial + syringe presentation
  Arms: Efgartigimod PH20 SC - vial + syringe

SUMMARY:
This is a randomized, open-label, parallel-group, single-dose study comparing the pharmacokinetics of efgartigimod in blood following a single administration of efgartigimod PH20 SC via a prefilled syringe versus a vial + syringe in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Is at least the local legal age of consent for participation in a clinical study and ≤55 years when signing the ICF
* Is capable of providing signed informed consent, and complying with protocol requirements
* Agrees to use contraceptive measures consistent with local regulations and the following: Women Of Child-Bearing Potential must have a negative serum hCG pregnancy test at screening and a negative urine hCG pregnancy test at baseline before receiving IMP.
* Has a BMI between 18 and 30 kg/m2 , inclusive, and a weight between 50 and 100 kg (inclusive) at screening

Exclusion Criteria:

* Has a known autoimmune disease or any medical condition that, in the investigator's judgment, would interfere with an accurate assessment of clinical symptoms or puts the participant at undue risk
* Has a history of malignancy, unless considered cured by adequate treatment with no evidence of recurrence for ≥3 years before the administration of IMP. Adequately-treated participants with the following cancers can be included at any time: Basal cell or squamous cell skin cancer; Carcinoma in situ of the cervix; Carcinoma in situ of the breast; Incidental histological findings of prostate cancer.
* Has a clinically significant active infection that is not sufficiently resolved in the investigator's opinion.
* Has a positive serum test at screening for active infection with any of the following: HBV indicative of an acute or chronic infection, unless associated with a negative HBsAg or negative HBV DNA test; HCV based on HCV antibody assay unless a negative RNA test is available ; HIV based on test results (regardless of therapy treatment or not).
* Has a clinically significant disease, recent major surgery (within 3 months of screening), or intends to have surgery during the study; or any other medical condition that, in the investigator's opinion, would confound the results of the study or put the participant at undue risk.
* Received a different IMP in another clinical study <12 weeks or 5 half-lives (whichever is longer) before screening.
* Is currently participating in another interventional clinical study. Has a known hypersensitivity to IMP or its excipients.
* Has abdominal skin condition that does not allow for absorption and assessment of local safety of the planned SC injection, as determined by the investigator.
* Has a history of (within 12 months before screening) or current alcohol, drug, or medication abuse, as assessed by the investigator.
* Is pregnant or lactating or intends to become pregnant during the study.
* Previously participated in an efgartigimod clinical study and received at least 1 dose of IMP.
* Is taking concomitant medications (except for oral contraceptives or occasional acetaminophen).
* Has a total IgG of <4 g/L at screening.
* Had a positive COVID-19 test result on day -1 or contact with someone with a known COVID-19 infection within 2 weeks before receiving IMP.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Primary PK parameters (Cmax) | Up to 29 days
  maximum observed plasma concentration
Primary PK parameters (AUC0-inf) | Up to 29 days
  area under the concentration-time curve from 0 to infinity

SECONDARY OUTCOMES:
Total IgG as percent change from baseline over time | up to 57 days
Total IgG as absolute change from baseline over time | up to 57 days
Safety parameters (number of AEs) | up to 85 days
Incidence of ADA against efgartigimod PH20 SC | up to 57 days
  Incidence of antidrug antibodies against efgartigimod PH20 SC
Second PK parameters (Tmax) | up to 57 days
  time to maximum concentration
Second PK parameters (AUC0-t) | up to 57 days
  area under the concentration-time curve from 0 to last quantifiable concentration
Second PK parameters (AUC0-168h) | up to 57 days
  area under the concentration-time curve from time 0 to168 hours
Second PK parameters (t1/2) | up to 57 days
  elimination half-life
Second PK parameters (Vz/F) | up to 57 days
  apparent volume of distribution
Second PK parameters (CL/F) | up to 57 days
  apparent clearance (total body clearance for extravascular administration divided by the fraction of dose absorbed, calculated using the observed value of the last nonzero concentration)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Investigator site 0010209, Tempe, Arizona
  - Investigator site 0010208, Lincoln, Nebraska

IPD SHARING:
Plan to Share IPD: Undecided